CLINICAL TRIAL: NCT05350436
Title: More Singing, Less Swinging - Is Singing Related to Improved Postural Control?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brunel University (Other)
Responsible Party: Principal Investigator, Adam Lewis, Lecturer in Physiotherapy, Brunel University
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 35423
Record Dates: First submitted 2022-03-30; First posted 2022-04-28 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Healthy Aging; Balance; Distorted; Singing
MeSH Terms: interventions — Singing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Young adult non singers (Experimental)
  Interventions: Behavioral: Balance Conditions; Behavioral: Singing
- Young adult singers (Experimental)
  Interventions: Behavioral: Balance Conditions; Behavioral: Singing
- Older adult non singers (Experimental)
  Interventions: Behavioral: Balance Conditions; Behavioral: Singing
- Older adult singers (Experimental)
  Interventions: Behavioral: Balance Conditions; Behavioral: Singing

INTERVENTIONS:
Behavioral: Balance Conditions — Balance Conditions: (~ 5 minutes in total)
  * Balance Condition 1 (Feet 20cm apart)
  * Balance Condition 2 (Feet together)
  * Balance Condition 3 (Tandem stance)
  Initial measurements of balance conditions serve two purposes: it generates a postural control baseline for us without the attribution of singing conditions, furthermore it allows us to separately measure long-term singing experience's effect on postural control, by assessing tasks differing in difficulty level. Balance conditions will be randomised to prevent a learning effect.
Behavioral: Singing — Singing Conditions: (~ 15 minutes)
  * Warmup - including jaw and breathing exercises
  * Singing Condition 1 (Spoken Happy Birthday - Traditional Tempo)
  * Singing Condition 2 (Sung Happy Birthday - Traditional Tempo
  * Singing Condition 3 (Spoken Happy Birthday - Fast Tempo)
  * Singing Condition 4 (Sung Happy Birthday - Fast Tempo)
  * Singing Condition 5 (Spoken Happy Birthday - Slow Tempo)
  * Singing Condition 6 (Sung Happy Birthday - Slow Tempo)
  Link to singing instructional video:
  https://www.dropbox.com/s/tro58i6vx6i6w3a/Singing%20Balance%20Exercise%20Video.mp4?dl=0
  Time stamps for the video:
  * Warmup (including jaw exercises and breathing exercises) - beginning at 2:55 until 6:06
  * Happy Birthday protocol - beginning at 15:26 until 20:21

SUMMARY:
This study will investigate the extent to which singing affects balance and breathing.

Singing therapy has potential as an adjunct or component of falls prevention programmes and in the treatment of breathing hypervigilance. Reducing fall risk, and levels of hypervigilance and anxiety could have widespread benefits on participants participation and quality of life.

Investigators will aim to recruit both singers and non singers from older and younger adult age groups. Investigators will then be able to determine the balance response in untrained healthy young adults to understand the affects of singing training and aging on balance. The participants' balance will be measured via a force plate as they perform a series of speaking and singing tasks. Other outcomes will include breathing specific anxiety and attention to breathing, and balance specific anxiety and attention to balance.

DETAILED DESCRIPTION:
Singing has become a popular arts-in-therapy activity used by physiotherapists as part of their clinical treatment. For example, Singing for Lung Health (SLH) programmes are used in the management of long-term respiratory conditions. These programmes involve group-based singing activities with a focus on breathing control and posture. There are indications that SLH is effective at alleviating symptoms of respiratory disease, likely due to a combination of physical, psychological and social mechanisms.

One main factor that could directly impact on breathing are affective and attentional changes. Reduced anxiety and depression through singing therapy has been suggested to improve breathing control and functioning in those with chronic respiratory conditions. Qualitative surveys have reported that participants find singing to be an "uplifting" activity and that singing with a group of peers may also help to combat isolation.

These changes may be accompanied by changes in allocation of attention. I.e., it is thought that anxiety leads to heightened vigilant monitoring of breathing, and that this hypervigilance leads to a switch in control of breathing from automatic to consciously processed, resulting in breathing dysfunction and breathlessness. Notably, normalisation of such excessive anxiety related vigilance may underpin the improvements that patients report after singing therapy, in terms of control of breathing and breathlessness during exacerbations. Singing therapy may therefore improve breathing control through reducing anxiety as well as associated attention to breathing. One aim of this study is to test this idea further, and to determine if singing impacts on breathing vigilance.

An additional potentially very important effect of singing interventions is that people may improve their balance control as well, both directly and indirectly. Breathing and postural control are tightly linked. We continuously need to make postural adjustment in response to disturbances due to (changes in) breathing - and especially so when breathing is effortful and accelerated. Several studies of SLH in patients with COPD report participants perceive singing had a positive impact on their posture. Also, recent studies suggest that expert singers have better postural control compared to novices. Better control over breathing thus may also improve postural control.

Indirectly, and similar to breathing vigilance, singing interventions may also help normalise individual's attention toward posture and balance. Fear of falling is common in people with respiratory conditions such as COPD. Typically, such fear / anxiety will lead to a strong, potentially excessive, increase in attention to balance. As with breathing, this "hypervigilance" can itself lead to distorted perception of unsteadiness. Singing therapy may therefore improve balance control through reducing anxiety and associated attention to movement.

Therefore, this study will also explore the effects of singing on balance control and associated changes in balance-related hypervigilance.

To investigate these questions, investigators planned a scoping study in which they:

* Aim to investigate the effects of singing on breathing control (e.g., breathing rate, breathing pattern assessment; see all outcomes below)
* Immediate: Effects of singing (varying demands) vs no-singing condition
* Long-term: differences between people with and without regular singing experience in terms of breathing control during no-singing vs singing conditions.
* Aim to investigate the effects of singing on breathing-related anxiety & vigilance (state anxiety, breathing vigilance; self-reported)
* Immediate effects (balance vs. balance + singing) & long-term effects (differences between groups with and without singing experience)
* Aim to investigate the effects of singing on balance control (sway, sway frequency)
* Immediate effects (balance vs. balance + singing) & long-term effects (differences between groups with and without singing experience)
* Aim to investigate the effects of singing on balance-related anxiety and vigilance (state anxiety, balance hypervigilance, conscious processing of balance; all self-reported)
* Again, immediate effects (balance vs. balance + singing) & long-term effects (differences between groups with and without singing experience)

ELIGIBILITY:
Inclusion Criteria:

* For young adults: 18 - 35 years of age
* For older adults: 60 years of age or older
* The "Older Adult" age group will be defined as adults aged 60 and older, based on the specifications of the World Health Organization (2017).
* The "Younger Adult" age group will be defined as adults aged 18 to 35 inclusive. There will be a buffer range of ages 36 to 59. This is being done to get a clear delineation between age groups.

Exclusion Criteria:

For all:

* Any respiratory, neurological, cardiac disease or deficit (and are on regular medication for it), and/or mobility issues.
* Have tested positive for COVID-19 in the last 15 days (van Kampen et al., 2021)
* Are diagnosed with Chronic COVID Syndrome
* Conditions limiting the ability to stand for >1 minute independently (e.g., chronic fatigue, recent injury affecting balance)
* Pregnancy (although this will not apply to older adults)
* Conditions limiting participating in singing activities (aphasia, dysarthria, dysphonia, speech impairments)

Investigating young adults allows to better isolate the effects of singing, as these individuals will not suffer from co-morbidities that may confound, modify or attenuate the effects. Conversely, the older adult group is relevant to study from a clinical point of view.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-02-25 (Actual); Primary Completion 2023-04-10 (Estimated); Study Completion 2023-04-10 (Estimated)

PRIMARY OUTCOMES:
Postural Sway Amplitude | 30 seconds during each balance condition 1
  An AMTI force plate (Optima AccuSway), will be used to measure postural sway this will be operationalised as "root-mean-square" sway signal throughout the trail (sample rate: 100Hz). Sway will be measured in both mediolateral and anterior-posterior directions
Postural Sway Amplitude | 30 seconds during each balance condition 2
  An AMTI force plate (Optima AccuSway), will be used to measure postural sway this will be operationalised as "root-mean-square" sway signal throughout the trail (sample rate: 100Hz). Sway will be measured in both mediolateral and anterior-posterior directions
Postural Sway Amplitude | 30 seconds during each balance condition 3
  An AMTI force plate (Optima AccuSway), will be used to measure postural sway this will be operationalised as "root-mean-square" sway signal throughout the trail (sample rate: 100Hz). Sway will be measured in both mediolateral and anterior-posterior directions
Postural Sway Amplitude | 30 seconds during each singing condition 1-6
  An AMTI force plate (Optima AccuSway), will be used to measure postural sway this will be operationalised as "root-mean-square" sway signal throughout the trail (sample rate: 100Hz). Sway will be measured in both mediolateral and anterior-posterior directions

SECONDARY OUTCOMES:
Sway frequency (in Hz) | 30 seconds during each balance condition 1
  sway frequency will be measured in both mediolateral and anterior-posterior directions
Sway frequency (in Hz) | 30 seconds during each balance condition 2
  sway frequency will be measured in both mediolateral and anterior-posterior directions
Sway frequency (in Hz) | 30 seconds during each balance condition 3
  sway frequency will be measured in both mediolateral and anterior-posterior directions
Sway frequency (in Hz) | 30 seconds during each singing conditions 1-6
  sway frequency will be measured in both mediolateral and anterior-posterior directions
Balance-Vigilance Questionnaire | Immediately after balance condition 1
  A balance vigilance questionnaire
Balance-Vigilance Questionnaire | Immediately after balance condition 2
  A balance vigilance questionnaire
Breathe-Vigilance Questionnaire | Immediately after balance condition 3
  A breathing vigilance questionnaire
Breathe-Vigilance Questionnaire | Immediately after each singing condition 1-6
  A breathing vigilance questionnaire
blood oxygen saturation (SpO2) | Immediately after balance condition 1
  oxygen saturation
blood oxygen saturation (SpO2) | Immediately after each singing condition 1-6
  oxygen saturation
Heart rate | immediately after balance condition 1
  heart rate
Heart rate | Immediately after each singing condition 1-6
  heart rate
Respiratory rate | Baseline measurement prior to all conditions for all participants
  breaths per minute
Respiratory rate | Immediately after balance condition 1
  breaths per minute
Respiratory rate | Immediately after each singing condition 1-6
  breaths per minute
Borg dyspnoea scale | Baseline assessment prior to all conditions for all participants
  participant completed measure of dyspnoea
Borg dyspnoea scale | Immediately after balance condition 1
  participant completed measure of dyspnoea
Borg dyspnoea scale | Immediately after balance condition 2
  participant completed measure of dyspnoea
Borg dyspnoea scale | Immediately after balance condition 3
  participant completed measure of dyspnoea
Borg dyspnoea scale | Immediately after each singing condition 1- 6
  participant completed measure of dyspnoea
Breathing Pattern Assessment Tool | Baseline measurement prior to conditions for all participants
  Researcher recorded observation of breathing pattern
Mental Readiness Form | Immediately after balance condition 1
  Measure of state anxiety
Mental Readiness Form | Immediately after balance condition 2
  Measure of state anxiety
Mental Readiness Form | Immediately after balance condition 3
  Measure of state anxiety
Mental Readiness Form | Immediately after each singing condition 1-6
  Measure of state anxiety
Timed Up and Go | Before any of the singing and balance conditions (baseline measurement (older adults))
  Measure of physical performance
Fall Efficacy Scale International | Before any of the singing and balance conditions a baseline measurement
  Patient reported outcome measure of risk of falls
State Trait Anxiety Inventory - Y2 | Baseline measurement prior to any condition for all participants
  Patient reported outcome measure of anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- Brunel University London Division of Physiotherapy, Uxbridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Other researchers can request access to data on reasonable request via email to the study investigators.

REFERENCES:
- [Background] Burdon JG, Juniper EF, Killian KJ, Hargreave FE, Campbell EJ. The perception of breathlessness in asthma. Am Rev Respir Dis. 1982 Nov;126(5):825-8. doi: 10.1164/arrd.1982.126.5.825. PMID 7149447
- [Background] Hodges PW, Gurfinkel VS, Brumagne S, Smith TC, Cordo PC. Coexistence of stability and mobility in postural control: evidence from postural compensation for respiration. Exp Brain Res. 2002 Jun;144(3):293-302. doi: 10.1007/s00221-002-1040-x. Epub 2002 Apr 13. PMID 12021811
- [Background] Lewis A, Cave P, Stern M, Welch L, Taylor K, Russell J, Doyle AM, Russell AM, McKee H, Clift S, Bott J, Hopkinson NS. Singing for Lung Health-a systematic review of the literature and consensus statement. NPJ Prim Care Respir Med. 2016 Dec 1;26:16080. doi: 10.1038/npjpcrm.2016.80. PMID 27906158
- [Background] Lord VM, Cave P, Hume VJ, Flude EJ, Evans A, Kelly JL, Polkey MI, Hopkinson NS. Singing teaching as a therapy for chronic respiratory disease--a randomised controlled trial and qualitative evaluation. BMC Pulm Med. 2010 Aug 3;10:41. doi: 10.1186/1471-2466-10-41. PMID 20682030
- [Background] Lord VM, Hume VJ, Kelly JL, Cave P, Silver J, Waldman M, White C, Smith C, Tanner R, Sanchez M, Man WD, Polkey MI, Hopkinson NS. Singing classes for chronic obstructive pulmonary disease: a randomized controlled trial. BMC Pulm Med. 2012 Nov 13;12:69. doi: 10.1186/1471-2466-12-69. PMID 23145504
- [Background] Oliveira CC, McGinley J, Lee AL, Irving LB, Denehy L. Fear of falling in people with chronic obstructive pulmonary disease. Respir Med. 2015 Apr;109(4):483-9. doi: 10.1016/j.rmed.2015.02.003. Epub 2015 Feb 14. PMID 25708268
- [Background] Peultier-Celli L, Audouin M, Beyaert C, Perrin P. Postural Control in Lyric Singers. J Voice. 2022 Jan;36(1):141.e11-141.e17. doi: 10.1016/j.jvoice.2020.04.019. Epub 2020 May 24. PMID 32456837
- [Background] Philip KE, Lewis A, Jeffery E, Buttery S, Cave P, Cristiano D, Lound A, Taylor K, Man WD, Fancourt D, Polkey MI, Hopkinson NS. Moving singing for lung health online in response to COVID-19: experience from a randomised controlled trial. BMJ Open Respir Res. 2020 Nov;7(1):e000737. doi: 10.1136/bmjresp-2020-000737. PMID 33239406
- [Background] Skingley, A. et al. 'Singing for Breathing': participants' perceptions of a group singing programme for people with COPD. Arts Health 6, 59-74 (2014).
- [Background] van Kampen JJA, van de Vijver DAMC, Fraaij PLA, Haagmans BL, Lamers MM, Okba N, van den Akker JPC, Endeman H, Gommers DAMPJ, Cornelissen JJ, Hoek RAS, van der Eerden MM, Hesselink DA, Metselaar HJ, Verbon A, de Steenwinkel JEM, Aron GI, van Gorp ECM, van Boheemen S, Voermans JC, Boucher CAB, Molenkamp R, Koopmans MPG, Geurtsvankessel C, van der Eijk AA. Duration and key determinants of infectious virus shedding in hospitalized patients with coronavirus disease-2019 (COVID-19). Nat Commun. 2021 Jan 11;12(1):267. doi: 10.1038/s41467-020-20568-4. PMID 33431879
- [Background] Vidotto LS, Bigliassi M, Jones MO, Harvey A, Carvalho CRF. Stop Thinking! I Can't! Do Attentional Mechanisms Underlie Primary Dysfunctional Breathing? Front Physiol. 2018 Jun 22;9:782. doi: 10.3389/fphys.2018.00782. eCollection 2018. No abstract available. PMID 29988475
- [Background] Vidotto LS, Carvalho CRF, Harvey A, Jones M. Dysfunctional breathing: what do we know? J Bras Pneumol. 2019 Feb 11;45(1):e20170347. doi: 10.1590/1806-3713/e20170347. PMID 30758427
- [Background] World Health Organisation (WHO) (2017). Mental Health of Older Adult. Available at: https://www.who.int/news-room/fact-sheets/detail/mental-health-of-older-adults. Accessed 17/01/22)
- [Background] World Health Organisation (WHO) (2021). Falls. Available at: https://www.who.int/news-room/fact-sheets/detail/falls (Accessed: 12/01/22)